CLINICAL TRIAL: NCT07209787
Title: A Prospective, Multicenter, Randomized Controlled Study Comparing Effect of Conventional Versus SIS-Reinforced Rectum Anastomosis On Anastomotic Leak Following Radical Resection of Mid-to-Low Rectal Cancer（SISReal）
Brief Title: SIS-Reinforced vs. Conventional Anastomosis for Mid-to-Low Rectal Cancer: A Multicenter RCT on Anastomotic Leak
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Beijing Chao Yang Hospital (Other)
Collaborators: Beijing Hospital (Other Government); Huashan Hospital (Other); First Affiliated Hospital of Gannan Medical University (Other); Guangdong Second Provincial General Hospital (Other); People's Hospital of Guangxi Zhuang Autonomous Region (Other); First Affiliated Hospital of Harbin Medical University (Other); Changhai Hospital, Naval Medical University (Unknown); Henan Provincial People's Hospital (Other); Hubei Cancer Hospital (Other); Hunan Provincial People's Hospital (Other); Tongji Hospital (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Second Hospital of Jilin University (Other); The Jiangxi Provincial People's Hospital (Unknown); The First Hospital of Lanzhou University, Gansu, China (Unknown); The First Affiliated Hospital of Nanchang University (Other); Nanjing Jiangning Hospital (Unknown); The First Affiliated Hospital of BaoTou Medical College (Other); The Affiliated Hospital of Qingdao University (Other); Qilu Hospital of Shandong University (Other); NORTHERN JIANGSU PEOPLE'S HOSPITAL 1900 (Unknown); Suzhou Municipal Hospital (Other); Taizhou People's Hospital (Unknown); First Affiliated Hospital of Wenzhou Medical University (Other); Zhongnan Hospital (Other); The Third Xiangya Hospital of Central South University (Other); First Affiliated Hospital of Xinjiang Medical University (Other); Yunnan Cancer Hospital (Other); The First Affiliated Hospital, Zhejiang University (Unknown); The First Affiliated Hospital of Zhengzhou University (Other); PLA Rocket Force Characteristic Medical Center (Other); The General Hospital of Western Theater Command (Other); China-Japan Friendship Hospital (Other); Sixth Affiliated Hospital, Sun Yat-sen University (Other); The Second Affiliated Hospital of Chongqing Medical University (Other); First Affiliated Hospital of Chongqing Medical University (Other); Zhoukou Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-科-689
Record Dates: First submitted 2025-09-29; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental)
  Interventions: Device: SIS-reinforced anastomosis
- control group (No Intervention)

INTERVENTIONS:
Device: SIS-reinforced anastomosis — This intervention uses a porcine small intestinal submucosa (SIS) reinforcement patch during rectal anastomosis. The sterile, biologic, acellular mesh is mounted onto the stapler anvil and cartridge. When fired, it encircles and externally reinforces the staple line. This provides immediate mechanical support and promotes healing by serving as a scaffold for tissue integration. It is a single-use, resorbable material intended to reduce anastomotic leakage by improving seal integrity, distinguishing it from standard unreinforced stapling or other synthetic/biologic grafts.
  Arms: Intervention arm

SUMMARY:
The goal of this clinical trial is to learn whether using a reinforcing material called SIS (small intestinal submucosa) during bowel connection after rectal cancer surgery can help prevent anastomotic leakage-a serious complication where the connection between two parts of the intestine fails to heal properly. This study will focus on patients with mid-to-low rectal cancer who are scheduled for surgery.

The main questions the study aims to answer are:

Does using an SIS-reinforced connection reduce the rate of anastomotic leakage within 30 days after surgery compared to standard connection methods?

Does it also reduce the need for a temporary stoma (an opening in the abdomen for waste removal)?

Researchers will compare two groups:

Intervention group: Patients who receive the SIS-reinforced connection during surgery.

Control group: Patients who receive the standard connection without reinforcement.

Participants in this study will:

Be randomly assigned to either the intervention or control group.

Undergo standard laparoscopic or robot-assisted rectal cancer surgery.

Be followed up at 30 days, 90 days, and 12 months after surgery to check for complications, stoma status, and quality of life.

This study is being conducted across multiple hospitals in China to ensure the results are reliable and widely applicable.

ELIGIBILITY:
Inclusion Criteria--

1. Age ≤ 85 years old, regardless of gender.
2. Patients with mid - low rectal cancer, where the lower edge of the cancer focus is ≤ 10 cm from the anus and who can undergo rectal anastomosis with a circular stapler (including mid - low and some ultra - low rectal anastomoses). This includes patients after neoadjuvant therapy, patients with insufficient function of important organs such as the heart, liver, and kidneys who can tolerate surgery, and patients after intestinal obstruction stent placement or chemotherapy after intestinal obstruction stent placement.
3. For patients who, after being fully informed by doctors, still clearly refuse neoadjuvant therapy (for advanced rectal cancer) and/or immunotherapy (for MSI - H/dMMR rectal cancer) and request direct surgery, they are generally not included in this study. If a patient insists on enrolling, the operating surgeon must have a second conversation with the patient and/or their family members, and sign in the medical record to confirm the following: The patient is aware of the existence of the neoadjuvant therapy/immunotherapy pathway but refuses the relevant treatment and insists on direct surgery. Only in this case can the patient be allowed to enroll.
4. Patients who received conversion therapy due to distant organ (such as liver, lung) metastasis before surgery and then underwent surgery with primary anastomosis can be included in this study. If organ metastasis is accidentally found during surgery, or if the small intestine or bladder in the pelvic floor is invaded, but the surgeon believes it does not affect rectal anastomosis, the patient does not need to withdraw from the study.
5. The patient or their authorized representative voluntarily signs the informed consent form and can cooperate to complete the follow - up during the trial.

Exclusion Criteria--

1. Patients who, through examination and pre - operative consultation, cannot tolerate routine surgery.
2. Patients who are currently participating in other clinical studies.
3. Since the test device (SIS reinforcement patch) is derived from porcine - sourced materials, out of respect for specific religious beliefs (such as Islam), we do not recommend that subjects whose beliefs prohibit contact with porcine - sourced products participate in this study. We will fully communicate this situation with all potential subjects, and the subjects will make their own decisions based on their personal beliefs and cultural backgrounds.
4. Patients who do not meet the NCCN and the National Health Commission of China's treatment standards for rectal cancer will not be included in this study. For example, patients who should receive neoadjuvant therapy before surgery should preferentially choose neoadjuvant therapy, and MSI - H/dMMR patients are required to undergo immunotherapy first.
5. Due to the possible difficulty in matching the number of patients/omissions with regular patients, patients who require lateral lymph node dissection and those who receive Ta - TME will not be included in this study.
6. Patients who, due to language or intellectual disabilities, cannot understand the content of the trial protocol, cannot complete the follow - up, or for whom the researcher deems there are other situations that are not suitable for enrollment (such as uncontrolled severe underlying diseases, mental illness, etc.).

Max Age: 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 966 (Estimated)
Dates: Start 2025-09-08 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Rate of anastomotic leak within 30 days post-surgery | From the date of surgery up to 30 days postoperatively
  Proportion of participants with an anastomotic leak (AL) within 30 days post-surgery. AL is a defect in the intestinal wall anastomosis, confirmed by clinical signs (e.g., fever, fecal drain output), imaging (CT scan with contrast extravasation or peri-anastomotic collections), or endoscopy. Leaks are graded per International Study Group of Rectal Cancer (ISREC) criteria: Grade A (no intervention), B (managed without reoperation), or C (requires reoperation).
Rate of anastomotic leak within 30 days post-surgery | From the date of surgery up to 30 days postoperatively.
  The proportion of participants experiencing an anastomotic leak (AL) within 30 days after surgery. AL is defined as a defect in the integrity of the intestinal wall at the anastomosis site, leading to communication between the intra- and extraluminal compartments. Diagnosis is based on a combination of clinical signs (e.g., fever, abdominal pain, fecal discharge from drain), imaging findings (extravasation of contrast on enema CT scan or presence of peri-anastomotic fluid/air collections), or endoscopic evidence. Leaks are graded per the International Study Group of Rectal Cancer (ISREC) classification: Grade A (requiring no active therapeutic intervention), Grade B (requiring active therapeutic intervention but manageable without reoperation), and Grade C (requiring reoperation).

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing chaoyang hospital, Beijing, Beijing Municipality, China